CLINICAL TRIAL: NCT01737346
Title: Phase 2 Clinical Trial of PC(Procarbazine-CCNU) Chemotherapy in Patients With Recurrent or Resistant Glioblastoma With Methylated MGMT
Brief Title: Procarbazine and Lomustine in Recurrent Glioblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Incheon St.Mary's Hospital (Other)
Collaborators: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Dong-Sup Chung, Professor, Department of Neurosurgery, Incheon St.Mary's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KNOG-1201
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Recurrent Glioblastoma Multiforme
Keywords: glioblastoma, recurrent, refractory, CCNU, procarbazine
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — Lomustine; Procarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lomustine and procarbazine (Experimental): 1 cycle (4 weeks) includes CCNU 75mg/m2 (D1) and procarbazine 60mg/m2 (D11-D24)by mouth for up to 6 cycles
  Interventions: Drug: lomustine and procarbazine

INTERVENTIONS:
Drug: lomustine and procarbazine — 1 cycle (4 weeks) includes CCNU 75mg/m2 (D1) and procarbazine 60mg/m2 (D11-D24)by mouth for up to 6 cycles
  Other Names: CCNU; Matulan

SUMMARY:
The combination therapy of temozolomide and radiation has been established as the standard therapy for the initial treatment of glioblastoma. However, the prognosis for patients with recurrent/ refractory glioblastoma is dismal, with a median survival of 3~6 months. There is no efficient and standard care at the time of recurrence or progression following temozolomide administration. Recently, many clinicians have reassessed the efficacy of second-line chemotherapeutic agents such as nitrosoureas for the treatment of recurrent/refractory glioblastoma. It is very important that the effect of the agent is sustained and the adverse effect is reduced to preserve the quality of life in recurrent settings. We have realized that the clinical features of Korean patients are very different from those of foreign patients. Therefore, it is mandatory to develop the new strategy for the treatment of Korean patients. We modify the PCV chemotherapy in the dose and administration schedule of CCNU and procarbazine to reduce the side effect, especially hematologic problems. The dose of CCNU is reduced to 75mg/m2 and the interval between CCNU and procarbazine is increased. Moreover, vincristine is excluded because BBB permeability of vincristine is very poor and the risk of neurotoxicity is high. We introduce the modified PC chemotherapy regimen for the treatment of recurrent/refractory glioblastoma, which is the first multicenter trial for glioblastoma patients in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or radiologically confirmed progressive or recurrent glioblastoma with methylated MGMT promoter
* Within 6 months after or during Stupp regimen (TMZ-RT CCRT + adjuvant TMZ), or After re-treatment of cyclic TMZ, 6 months later after Stupp regimen
* KPS ≥ 60%
* Age ≥ 20 years
* At least two weeks apart from prior surgery and prior chemotherapy
* Adequate hematologic, liver, and renal functions
* Unstained slides for central pathology review
* Signed informed consent

Exclusion Criteria:

* Prior malignancy within 5 years except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and carcinoma in situ of the cervix
* maternity or breastfeeding
* Evidence of active infection within 2 weeks prior to study
* Previous treatment with procarbazine and/or CCNU
* Evidence of leptomeningeal metastasis
* Unable to comply with the study protocol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-09 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
6-month progression free survival | March 31, 2014

CONTACTS AND LOCATIONS:
Overall Officials: Don-Sup Chung, MD, Principal Investigator — Incheon St. Mary Hispital
Locations (1):
- Ajou University Hospital, Wonchondong, Suwon, South Korea